CLINICAL TRIAL: NCT04770363
Title: Comparison Between the Effect of Unihemispheric and Bihemispheric Transcranial Direct Current Stimulation on Spasticity and Motor Outcome in Subacute Ischemic Stroke Patients: as Add on Therapy
Brief Title: Comparison Between Unihemispheric and Bihemispheric TCDS in Subacute Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0106522
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic; Stroke, Acute; Stroke, Lacunar; Hemiparesis; Hemiplegia; Motor Activity; Spastic; Spasticity, Muscle; Hemiplegic Gait
MeSH Terms: conditions — Ischemic Stroke; Stroke; Stroke, Lacunar; Paresis; Hemiplegia; Motor Activity; Muscle Spasticity; Gait Disorders, Neurologic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will participate into the study, each patient will undergo a detailed neurological examination through filling out a medical sheet questionnaire and checking the most common risk factors of stroke and other parameters. ActivaDose tDCS (USA), the only FDA cleared device available for tDCS will be used in the clinical study. Thirty patients will be allocated randomly into three group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) To make sure that no bias should enter the assessment of the results, neither the patient nor the external assessor will be aware whether active tDCS will be applicated to a particular case. The patients don't know if which group they are participated in, bihemispheric, unihemispheric, of sham group, external assessor was recruited to assess patients after the intervention ended.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Bihemispheric Stimulation Group (Experimental): The first group tDCS bihemispheric stimulation consisted of 20 minutes of 2 mA direct current with the anode placed over the ipsilesional and the cathode over the contralesional motor cortex M1 (C3 and C4 of the international 10 -20 EEG electrode system).
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Unihemispheric Stimulation Group (Experimental): The second group unilateral stimulation, the anode placed over the ipsilesional motor cortex M1 (C3 or C4 of the international 10 -20 EEG electrode system) and the cathode over contralesional supraorbital bone.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham Group (Sham Comparator): The third sham group, the anode placed over the ipsilesional motor cortex M1 (C3 or C4 of the international 10 -20 EEG electrode system) and the cathode over contralesional supraorbital bone, but delivering no current.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is an emerging non-invasive brain stimulation technique which has been utilized in examining cortical function in healthy subjects and also showed significant outcome in neurological rehabilitation. A safe, portable, noninvasive painless, reversible, selective and focal brain stimulation technique, applied by sponge electrodes over the scalp. tDCS is capable of modulating the excitability of targeted brain zones through delivering a sustained direct current (DC), showed altering neuronal membrane potentials based on the polarity of the current. Researchers demonstrated modulating effects of anodal (increases cortical excitability) and cathodal (decreases cortical excitability) tDCS on brain tissue. The expected effects of tDCS brain stimulation exceeds the duration. Animal studies showed neuronal depolarization and increasing neuronal excitability of the anodal stimulation, and opposite results with cathodal stimulation.
  Other Names: (tDCS)

SUMMARY:
This is a randomized clinical trial to study the effect of tDCS in participants with subacute ischemic stroke, the study participants will be randomly assigned into three groups; bihemispheric, unihemispheric and sham group.

DETAILED DESCRIPTION:
Despite the central origin of stroke affecting the primary motor cortex M1, majority of the rehabilitative techniques of physical therapy and occupational therapy practice depending peripheral methods for gaining motor functions. There is a great need to develop methods in order to improve the outcome of physical or medical rehabilitation and enhance long-term functional outcome. Many researches' work over the past several years have inspected the use of transcranial direct current stimulation (tDCS) to promote the advantageous effect of neurological rehabilitation.

The aim of This study Is to compare between the effect of unihemispheric and bihemispheric tDCS on the motor outcome, and spasticity in sub-acute ischemic stroke patients.

Thirty sub-acute ischemic stroke patients participated in the study, randomly assigned to one of three groups-tDCS bihemispheric or unihemispheric or sham group. Those patients had stroke in the last 3 months at maximum with NIH stroke score less than 25. ActivaDose tDCS (USA), the only FDA cleared device available for tDCS used in the clinical study to deliver noninvasive brain stimulation, consisted of 20 minutes of 2 mA in each session for twelve sessions three sessions per week. All participants received physiotherapy and rehabilitation therapy was tailored to meet all patients' deficits, and lasted a total of 45 minutes per day, 3 days per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those patients had stroke in the last 3-6 months.
* Subcortical stroke of middle cerebral artery (MCA), caused unilateral hemiplegia.
* National institute of health stroke scale (NIHSS) motor deficits section with score 2 to 15.

Exclusion Criteria:

* Patient with second onset of stroke or history of Transient ischemic attack (TIA)
* Metallic Implant or heart pacemakers.
* Primary cerebral or subarachnoid hemorrhagic stroke.
* Seizure or epilepsy or history of epilepsy at the family.
* Intracranial abscess or brain tumor.
* Cardiovascular disease myocardial infarction, heart failure (unstable cardiac status).
* Atrial Fibrillation or paroxysmal AF in the last 30 days.
* Congenital heart diseases.
* Presence of any other neurological or psychiatric disorder.
* Cognitive/consciousness disorders.
* Oher conditions should be excluded (e.g. tumor, cancer, rheumatologic, Lung disease related to infection, renal/ hepatic diseases, deep venous thrombosis and autoimmune diseases).
* Speech disorders (Dysarthria & Aphasia).
* NIH Stroke score above 25, will be excluded.
* Patients who underwent thrombolytic therapy or any vascular interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | 1 Month
  To assess the upper and lower extremities, motor and sensory recovery assessment.
  Maximal attainable score is 226, means a good and functional physical state.
Modified Ashworth Scale (MAS) | 1 Month
  To assess the spasticity within the upper and lower extremities, score ranges from 0-4 with 5 choices. 0 indicates no resistance and 4 indicates rigidity. Higher scores indicate worse outcome.
Brain-Derived Neurotrophic Factor (BDNF) concentration | 1 Month
  is assessed pre and post-treatment for all of the participants using (ELISA) molecular test, the difference between pre and post-treatment will be only assessed, no normal range is quantified.

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale, NIH Stroke Scale (NIHSS) | Assessed for one time during participant recruitment
  to objectively assess the impairment caused by a stroke, score ranges from 0-42. Higher scores indicate worse outcome and severity. 0 is normal state of any participant.
Berg Balance Scale | 1 Month
  To assess the body balance and rısk of fall within the upper and lower extremities, The test is scored using a 5-point ordinal scale (0-4) with detailed descriptors for each score. 0 indicates inability to obtain the task and 4 ability to fully obtain the task. Higher scores indicate good outcome. The total score ranges from 0 to 56.

CONTACTS AND LOCATIONS:
Overall Officials: Nema Mohamed, PHD Prof, Principal Investigator — Faculty of Science - Alexandria University
Locations (1):
- Ethics Committee - Alexandria Faculty of Medicine, Alexandria, Egypt